CLINICAL TRIAL: NCT00417248
Title: A Phase II Trial of Concurrent Cisplatin/Etoposide/Radiotherapy Followed by Consolidation Sorafenib in Patients With Inoperable Stage III Non-Small Cell Lung Cancer (NSCLC): Hoosier Oncology Group LUN06-107
Brief Title: Cisplatin/Etoposide/Radiotherapy Followed by Consolidation Sorafenib for Inoperable Stage III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Negative sorafenib results from ESCAPE trial and safety concerns of regimen
Sponsor: Nasser Hanna, M.D. (Other)
Collaborators: Bayer (Industry); Amgen (Industry); Walther Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Nasser Hanna, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG LUN06-107
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; Radiotherapy; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational Treatment (Experimental): Cisplatin/Etoposide/Radiotherapy followed by Sorafenib in patients with inoperable stage III non-small cell lung cancer
  Interventions: Drug: Cisplatin; Drug: Etoposide; Procedure: Radiotherapy; Drug: Sorafenib

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 50 mg/m2 IV, days 1 and 8 of 28 day cycle
Drug: Etoposide — Etoposide 50 mg/m2 IV, days 1-5 of 28 day cycle
Procedure: Radiotherapy — Concurrent chest radiation (planned dose is 5940 cGy with an additional, optional boost of 1080 cGy to a total allowed dose of 7020 cGy)
Drug: Sorafenib — Maintenance therapy of Sorafenib 400 mg PO BID, to begin a minimum of 6 and maximum of 9 weeks from completion of chemo-radiotherapy until PD, intolerable toxicity, or up to 6 months

SUMMARY:
Sorafenib has demonstrated in vivo anti-tumor efficacy. This trial will evaluate the safety and preliminary efficacy of sorafenib following chemoradiation in locally advanced NSCLC.

DETAILED DESCRIPTION:
Outline: This is a multi-center study.

Chemotherapy/radiation therapy (2 cycles)

* Cisplatin 50 mg/m2 IV days 1 and 8 of 28 day cycle
* Etoposide 50 mg/m2 IV days 1-5 of 28 day cycle
* Concurrent chest radiation (planned dose is 5940 cGy with an additional, optional boost of 1080 cGy to a total allowed dose of 7020 cGy) with the following:

Maintenance therapy of Sorafenib 400 mg PO BID of 28 day cycle, to begin a minimum of 6 and maximum of 9 weeks from completion of chemo-radiotherapy until PD, intolerable toxicity, or up to 1 year.

Patients with progressive disease will discontinue treatment.

ECOG performance status 0 or 1

Hematopoietic:

* Absolute neutrophil count (ANC) ≥ 1500 mm3
* Platelet count ≥ 100,000 mm3
* Hemoglobin ≥ 9 g/dL
* PT or INR < 1.5 x ULN unless on anti-coagulant therapy
* PTT < 1.5 x ULN unless on anti-coagulant therapy

Hepatic:

* Bilirubin ≤ 1.5 x ULN
* ALT ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement)
* AST ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement)

Renal:

* Creatinine < 1.5 X upper limit of normal (ULN)

Cardiovascular:

* No significant history of cardiac disease: Congestive heart failure > class II NYHA.
* Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within 90 days prior to registration for initial therapy) or myocardial infarction within 6 months prior to registration for initial therapy.

Respiratory:

* FEV1 ≥ 1 liter by spirometry within 60 days prior to registration for initial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of non-small cell lung cancer (NSCLC).
* Measurable or non-measurable disease per RECIST.
* Unresectable Stage IIIA or IIIB disease as evaluated by imaging.
* Must be age ≥ 18 years at the time of consent.
* Written informed consent and HIPAA authorization for release of personal health information.
* Females of childbearing potential and males must be willing to use an effective method of contraception.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for initial therapy.

Exclusion Criteria:

* No prior chemotherapy or radiotherapy for lung cancer.
* No positive supraclavicular or scalene lymph nodes extending up into the cervical region.
* No superior sulcus (pancoast tumors).
* No malignant pleural effusions. The only exception is a patient with a pleural effusion visible only on CT scan (and not visible on CXR) OR deemed too small to tap.
* No clinically significant or malignant pericardial effusions.
* No CNS metastases.
* No unintended weight loss (> 5% body weight) in the preceding 90 days prior to registration for initial therapy.
* No treatment with any investigational agent within 30 days prior to being registered for initial therapy.
* No prior therapy with a Ras pathway inhibitor or anti-angiogenic agent.
* No other active cancers.
* Females must not be breastfeeding.
* No active clinically serious infections as judged by the treating investigator (> CTC v3, Grade 2) including known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* No major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration for initial therapy.
* No anticipation of need for major surgical procedure during the course of the study.
* No minor surgical procedures such as fine needle aspirations or cone biopsies within 7 days prior to registration for initial therapy.
* No history of allergic reactions to drugs utilizing the vehicle polysorbate 80 + polyethylene glycol (etoposide).
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to registration for initial therapy.
* No use inhibitors or inducers of the cytochrome p450 system CYP3A4 enzyme or other medications such as aprepitant, ketoconazole, itraconazole, quinidine, digoxin, cyclosporine, ritonavir, grapefruit products, St. John's Wort, rifampin (rifampicin), carbamazepine, phenytoin, dexamethasone, and phenobarbital.
* No evidence or history of bleeding diathesis or coagulopathy.
* No serious non-healing wound, ulcer, or bone fracture.
* No known or suspected allergy to sorafenib.
* No uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management.
* No thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within 6 months prior to registration for initial therapy.
* No pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks prior to registration for initial therapy.
* No hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to registration for initial therapy.
* No condition that impairs patient's ability to swallow whole pills or any malabsorption problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (8):
- United States (8):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Oncology Partners Network, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin/Etoposide/Radiotherapy Followed by Sorafenib: Cisplatin/Etoposide/Radiotherapy followed by Sorafenib in patients with inoperable stage III non-small cell lung cancer
  Cisplatin: Cisplatin 50 mg/m2 IV, days 1 and 8 of 28 day cycle
  Etoposide: Etoposide 50 mg/m2 IV, days 1-5 of 28 day cycle
  Radiotherapy: Concurrent chest radiation (planned dose is 5940 cGy with an additional, optional boost of 1080 cGy to a total allowed dose of 7020 cGy)
  Sorafenib: Maintenance therapy of Sorafenib 400 mg PO BID, to begin a minimum of 6 and maximum of 9 weeks from completion of chemo-radiotherapy until PD, intolerable toxicity, or up to 6 months
Period: Overall Study
Arm/Group | Cisplatin/Etoposide/Radiotherapy Followed by Sorafenib
Started | 8
Completed | 0
Not Completed | 8
Not completed — Study Terminated | 6
Not completed — Death | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin/Etoposide/Radiotherapy Followed by Sorafenib
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: Years] | 66.50 [59 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression (TTP)
Time Frame: 18 months
Population: The primary objective for this study was not analyzed due to termination of the study. No participants were on-study for a sufficient period of time to collect or analyze the time to disease progression data.
Arm/Group | Cisplatin/Etoposide/Radiotherapy Followed by Sorafenib
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Time Frame: 18 months
Population: Data for this outcome measure was not collected or analyzed due to the early termination of the study.
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Duration of OnStudy time, up to two 28 day cycles.
Arm/Group | Cisplatin/Etoposide/Radiotherapy Followed by Sorafenib
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin/Etoposide/Radiotherapy Followed by Sorafenib (N=8)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin/Etoposide/Radiotherapy Followed by Sorafenib (N=8)
ALKALINE PHOSPHATASE (Investigations) | 1 (2)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 1 (1)
ALLERGY/IMMUNOLOGY - OTHER (Immune system disorders) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 5 (5)
CONSTIPATION (Gastrointestinal disorders) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4)
CREATININE (Investigations) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 3 (4)
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 5 (6)
EDEMA: LIMB (Blood and lymphatic system disorders) | 1 (1)
ESOPHAGITIS (Gastrointestinal disorders) | 3 (4)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 6 (8)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
HEMOGLOBIN (Blood and lymphatic system disorders) | 3 (7)
HEMORRHAGE/BLEEDING - OTHER (General disorders) | 1 (1)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOT FLASHES/FLUSHES (Endocrine disorders) | 1 (1)
INSOMNIA (General disorders) | 1 (1)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 2 (2)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ESOPHAGUS (Gastrointestinal disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTRAOCULAR (Eye disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (5)
NEUROPATHY: MOTOR (Nervous system disorders) | 2 (2)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / ESOPHAGUS (Gastrointestinal disorders) | 3 (3)
PAIN / HEAD/HEADACHE (General disorders) | 1 (1)
PAIN / THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 2 (3)
SYNCOPE (FAINTING) (Nervous system disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (4)
WEIGHT LOSS (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No